CLINICAL TRIAL: NCT04853927
Title: Proxalutamide Treatment for COVID-19 Patients in Intensive Care Unit
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor to focus on hospitalised patients
Sponsor: Applied Biology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KP-DRUG-SARS-004
Record Dates: First submitted 2021-04-17; First posted 2021-04-22 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-02

CONDITIONS: Covid19; SARS (Severe Acute Respiratory Syndrome)
Keywords: Proxalutamide; Androgen; Anti-androgen
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — proxalutamide

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective, interventional, placebo controlled, double-blinded, randomized parallel assignment study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proxalutamide + Standard of Care (Active Comparator): Proxalutamide + standard of care as determined by the PI
  Interventions: Drug: Proxalutamide
- Placebo + Standard Care (Placebo Comparator): Placebo + Standard of care as determined by the PI
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Proxalutamide — Proxalutamide 300mg q.d suspension
  Arms: Proxalutamide + Standard of Care
Drug: Placebo — Proxalutamide 300mg q.d placebo
  Arms: Placebo + Standard Care

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Proxalutamide as a treatment for COVID-19 patients in the intensive care unit

DETAILED DESCRIPTION:
During the continuing SARS-CoV-2 (COVID-19) pandemic, several studies have reported a significant difference in the rate of severe cases between adult females and adult males (42% vs 58%). Among children under the age of 14, the rate of severe cases was reported to be extremely low. To explain this difference, several theories have been proposed including cigarette smoking and lifestyle habits. However, no theory fits both the gender difference in severe cases as well as reduced risk in pre-pubescent children. Our past research on male androgenetic alopecia (AGA) has led us to investigate an association between androgens and COVID-19 pathogenesis. In normal subjects, androgen expression demonstrates significant variation between men and women as well as between adults and pre-pubescent children.

SARS-CoV-2 primarily infects type II pneumocytes in the human lung. SARS-CoV-2 enters pneumocytes, by anchoring to the ACE2 cell surface receptor. Prior to receptor binding, viral spike proteins undergo proteolytic priming by the transmembrane protease, serine 2 (TMPRSS2). TMPRSS2 inhibition or knock down reduces ability of SARS-CoV-1 (a related virus to SARS-CoV-2) to infect cells in vitro.Additionally, TMPRSS2 also facilitates entry of influenza A and influenza B into primary human airway cells and type II pneumocytes.

The human TMPRSS2 gene has a 15 bp androgen response element and in humans, androgens are the only known transcription promoters for the TMPRSS2 gene. In a study of androgen-stimulated prostate cancer cells (LNCaP), TMPRSS2 mRNA expression increase was mediated by the androgen receptor. Further, the ACE2 receptor, also critical for SARS-CoV-2 viral infectivity, is affected by male sex hormones with higher activity found in males.

Previously, the investigators have reported the results from two retrospective cohort analysis demonstrating the protective effect of 5-alpha-reductase inhibitors (5ARi) for men with COVID-19. In a study of 77 men hospitalized with COVID-19 the investigators found among men taking 5ARis, 8% were admitted to the ICU compared to 58% of men not taking 5ARis (P = 0.0015). In the cohort, 5ARis were associated with reduced risk for ICU admissions RR 0.14 (95% CI: 0.02-0.94).Similarly, the investigators have demonstrated that the frequency of COVID-19 symptoms was drastically reduced for men using 5ARis in an outpatient setting. A statistically significant (p<0.05) reduction in the frequency of 20 of the 29 clinical symptoms was observed in AGA men using 5ARis compared to AGA men not using 5ARis. For example, 38% and 2% of men presented with low-grade fever, 60% and 6% with dry cough, and 88% and 15% reported anosmia in the non-5ARi and 5ARi groups, respectively.18

One limitation of 5ARis is the time course required to achieve systemic DHT reductions. As such, the investigators explored the use of a novel second generation androgen receptor antagonist Proxalutamide as a means for rapid reduction in AR activity. Proxalutamide (GT0918) demonstrates a dual mechanism of action. It is highly effective in inhibiting AR as well as exhibiting pharmacological effects of inducing the down-regulation of AR expression; the mechanism that is not present in bicalutamide and enzalutamide. Because of the dual mechanism of action, it is expected to be a more effective and less toxic second-generation anti-androgen drug therapy. Clinical evidence has demonstrated that Proxalutamide lowers AR expression and activity. Additionally, it has been reported that Proxalutamide lowers the expression of ACE2. Both would be beneficial for preventing SARS-CoV-2 entry into lung cells. In addition, none of the 5ARis currently approved by the US FDA have been tested in phase I studies in women. As such, thet are not recommended for women. Phase I studies for Proxalutamide have been successfully completed in both men and women.

In December 2020, the investigators completed a double-blinded, randomized, prospective, investigational study of Proxalutamide Treatment for Non-Hospitalized COVID-19 Male Patients (NCT04446429). The length of the study was 30 days. Proxalutamide was administered 200mg q.d. for 15 days. Men enrolled in the study were 50 years and older. Two hundred and sixty two men completed the study. 134 men were assigned to the Proxalutamide group and 128 men were assigned to the control group. Thirty five subjects were hospitalized in the control group compared to zero in the Proxalutamide group. The proportion of COVID-19 patients hospitalized was significantly different between the Proxalutamide and control arms; χ2 (1) = 42.051, p<.0001. The difference in proportions was 27.30% with a 95%CI: [19.79%, 35.59%]. No subject receiving Proxalutamide died compared to 2 (1.56%) in the control group. There were no treatment related adverse event reported during the course of the study.

Based on the results of the Proxalutamide Treatment for Non-Hospitalized COVID-19 Male Patients study (NCT04446429), the purpose of this study is to assess the efficacy and safety of Proxalutamide as a treatment for COVID-19 patients in the intensive care unit

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to the hospital with symptoms of COVID-19
2. Male and females age ≥18 years old
3. Laboratory confirmed positive SARS-CoV-2 rtPCR test within 14 days prior to randomization or confirmed lung involvement by CT scan
4. Clinical status on the COVID-19 Ordinal Scale of 6 or 7
5. Coagulation: INR ≤ 1.5×ULN, and APTT ≤ 1.5×ULN
6. Subject (or legally authorized representative) gives written informed consent prior to performing any study procedures
7. Subject (or legally authorized representative) agree that subject will not participate in another COVID-19 trial while participating in this study

Exclusion Criteria:

1. Subject enrolled in a study to investigate a treatment for COVID-19
2. Subject taking an anti-androgen of any type including: androgen depravation therapy, 5-alpha reductase inhibitors, etc…
3. Patients who are allergic to the investigational product or similar drugs (or any excipients);
4. Subjects who have malignant tumors in the past 5 years, with the exception of completed resected basal cell and squamous cell skin cancer and completely resected carcinoma in situ of any type
5. Subjects with known serious cardiovascular diseases, congenital long QT syndrome, torsade de pointes, myocardial infarction in the past 6 months, or arterial thrombosis, or unstable angina pectoris, or congestive heart failure which is classified as New York Heart Association (NYHA) class 3 or higher, or left ventricular ejection fraction (LVEF) < 50%, QTcF > 450 ms
6. Subjects with uncontrolled medical conditions that could compromise participation in the study(e.g. uncontrolled hypertension, hypothyroidism, diabetes mellitus)
7. Known diagnosis of human immunodeficiency virus(HIV) , hepatitis C, active hepatitis B, treponema pallidum (testing is not mandatory）
8. Alanine Transaminase (ALT) or Aspartate Transaminase (AST) > 5 times the upper limit of normal.
9. Estimated glomerular filtration rate (eGFR) < 30 ml/min
10. Severe kidney disease requiring dialysis
11. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective contraception, as shown below, throughout the study and for 3 months after stopping GT0918 treatment. Highly effective contraception methods include:

    * Total Abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception, or
    * Use of one of the following combinations (a+b or a+c or b+c):

      1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception.
      2. Placement of an intrauterine device (IUD) or intrauterine system (IUS) ;
      3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository ;
    * Female sterilization (have had prior surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment ;
    * Male sterilization (at least 6 months prior to screening). For female patients on the study, the vasectomized male partner should be the sole partner for that patient;
    * In case of use of oral contraception women should have been stable for a minimum of 3 months before taking study treatment. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment, is she considered not of child bearing potential;
12. Sexually active males must use a condom during intercourse while taking the drug and for 3 months after stopping GT0918 treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid
13. Subject likely to transfer to another hospital within the next 28 days
14. Subject (or legally authorized representative) not willing or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of death | Day 28
  Defined as the number of subjects who have died in each arm divided by the number of subjects randomized to the treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fonseca, MD, Principal Investigator — Samel Hospital; Flavio Cadegiani, MD, Principal Investigator — Corpometria
Locations (1):
- Samel Hospital, Manaus, Amazonas, Brazil